CLINICAL TRIAL: NCT04392466
Title: Comparison of Cognitive and Motor Dual Task Gait Characteristics in Individuals With Transtibial, Transfemoral Amputation and Healty Individuals
Brief Title: Comparison of Dual Task Gait Characteristics in Individuals With Amputation and Healty Individuals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Senem Demirdel, PhD, Pricipal Investigator, Hacettepe University
Other Study IDs: GO 20/23
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Dual Task; Amputation; Gait

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Transtibial amputees: People who use transtibial prosthesis.
  Interventions: Other: walking on the treadmill
- Transfemoral amputees: People who use transfemoral prosthesis.
  Interventions: Other: walking on the treadmill
- Healty individuals: Healty individuals
  Interventions: Other: walking on the treadmill

INTERVENTIONS:
Other: walking on the treadmill — Participants will walk on the treadmill under single task, cognitive dual task and motor dual task conditions.

SUMMARY:
In amputee, dual task has been found to cause a decrease in walking speed. However, there is no study of how gait characteristics are affected when the speed does not change. The aim of this study is to compare the time-distance characteristics of walking with single task, cognitive dual task, motor dual task in transtibial, transfemoral amputee and healthy people.

DETAILED DESCRIPTION:
Walking is a complex task in which sensory and cognitive systems must be involved. The lower extremity amputee may need to use cognitive resources to focus on walking, monitor and control the prosthetic movements. The need to use cognitive resources may be higher in those with more proximal level amputation, such as above-knee level. The role of cognition and concentration is revealed by a cognitive task performed with posture and gait control using the dual task method. The dual task paradigm provides information about the automation of the default processes that underpin good performance disclosure. This approach involves performing two tasks at the same time. Dual task is divided into primary task and secondary task. The performance of the primary task while performing a single task is recorded. If there is a drop in performance when the secondary task is added, this indicates that the primary task needs high attention.

In proximal amputations, with the lost of movement system structures, functional impairment increases. Amputation from the proximal level affects daily life activities and walking ability more. Above-knee amputees reported more functional difficulties in ambulatory ambulation than transtibial amputee.

The aim of this study is to compare the time-distance characteristics of walking with single task, cognitive dual task, motor dual task in transtibial, transfemoral amputee and healthy people.

ELIGIBILITY:
Inclusion Criteria:

* Using a transtibial or transfemoral prosthesis for at least 1 year,
* Between the ages of 18-65,

Exclusion Criteria:

* To be diagnosed as a neurological, orthopedic, cognitive disorder,
* Having a condition other than amputation that may affect gait.
* Having different permanent disabilities other than amputation,
* Using walking aid,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Transtibial amputees, Transfemoral amputees, Healty individuals
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-06-12 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Walking speed | Two minutes
  Distance per second
Coefficient of variation | Two minutes
  Stride length variability coefficient

SECONDARY OUTCOMES:
Step length | Two minutes
  Length of right and left steps in cm
Time on each foot | Two minutes
  The period on right foot and left foot
Average step cycle | Two minutes
  Yhe period of step cycle

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Erbahçeci, Prof, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepeu, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demirdel S, Erbahceci F, Yazicioglu G. The effects of cognitive versus motor concurrent task on gait in individuals with transtibial amputation, transfemoral amputation and in a healthy control group. Gait Posture. 2022 Jan;91:223-228. doi: 10.1016/j.gaitpost.2021.10.036. Epub 2021 Oct 27. PMID 34741932